CLINICAL TRIAL: NCT04799119
Title: The Evaluation of a Multi-site Imitation Based Animal Assisted Intervention for Children With Developmental Disabilities and Their Family Dog
Brief Title: Multi-site Animal Assisted Intervention for Children With DD and Their Family Dog
Acronym: DAID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Megan MacDonald, Professor, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-0816
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Physical Activity; Social Wellbeing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized control trial experimental/treatment group and control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAID dog training (Experimental): 'Do As I Do' (DAID) dog training employs operant conditioning to train dogs to copy the behavior of their owner upon hearing the verbal cue 'Do it', similar to teaching a dog the rules behind the game 'Simon Says'. Once this rule has been established and generalized, something that can be achieved in dogs by practicing with only 3-6 initially learned behaviors, owners can demonstrate new actions and use the cue 'Do it' to prompt a matched, imitative, behavioral response.
  Interventions: Behavioral: Do As I Do (DAID) dog training
- Control (No Intervention): No intervention (waitlisted and will be provided with the experimental condition post-study completion).

INTERVENTIONS:
Behavioral: Do As I Do (DAID) dog training — Children and their family dog will participate in this dog training program.
  Arms: DAID dog training

SUMMARY:
The study purpose is to evaluate a novel multidisciplinary approach to fostering a therapeutic partnership between the participants with developmental disabilities and the participants family dog. This will culminate in an Animal Assisted Intervention aimed at increasing activity levels, enhancing social support, and increasing feeling of responsibility and wellbeing within this population.

DETAILED DESCRIPTION:
The goal of this proposal is to evaluate a large scale novel multidisciplinary approach to fostering atherapeutic partnership between adolescents with developmental disabilities (DD) and the participants family dog. The investigators will evaluate imitative 'Do As I Do' (DAID) training into a unique Animal Assisted Intervention (AAI) aimed at increasing activity levels, enhancing social support by promoting a stronger dog-human bond, and increasing feelings of responsibility and wellbeing within this population.

The investigators propose to address the critical need for empirical evaluation of novel theoretically based multi-site animal assisted interventions through the following specific aims.

Specific Aim 1: To evaluate a novel multi-site DAID dog training intervention to promote physical activity in adolescents with developmental disabilities.

Specific Aim 2: To evaluate the impact of a multi-site DAID intervention on the adolescent's quality of life and feelings of social wellbeing.

Specific Aim 3: To evaluate the impact of a multi-site DAID intervention on the child-dog relationship and mutual wellbeing.

Participant Population: Adolescent participants with a developmental disability, between the ages of 10-17 years will be recruited through community-based programs/organizations associated with children with DDs in around our sites. A DD will be confirmed through parent report (e.g., initial recruitment conversations, and documented through the initial demographic questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Age 10-17 years
* Developmental disability (per parental report)
* Possesses family dog
* Participant can follow basis instructions.

Exclusion Criteria:

* Cannot follow basic instructions.
* Non english-speakers.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | One year
  Physical activity will be measure through accelerometry.

SECONDARY OUTCOMES:
Social well-being | One year
  Pediatric Quality of Life Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Megan MacDonald, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Due to the age range of the participants and targeted sample of children with disabilities as well as the small sample size (N=100), data will not be uploaded to NIH sharing tools.